CLINICAL TRIAL: NCT06179576
Title: Connect to Baby: A Pilot Study of a Parenting and Coparenting Program for New Parents
Brief Title: Connect to Baby: A Pilot Study of a Parenting and Coparenting Program
Acronym: CTB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Rebecca Ryan, Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21HD108499 (NIH)
Record Dates: First submitted 2023-05-18; First posted 2023-12-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Parenting
Keywords: Parent Education

STUDY DESIGN:
Intervention Model Description: Dyads in the EHS-CTB hybrid condition will receive 6 individual sessions of CTB conducted by trained facilitators. The first session would be at the center, the 2nd through 5th would be remote, and 6th would be at the EHS center as a group session with other families. Sessions will occur approximately one to two weeks apart, allowing for program completion within 10 weeks. During the first in-person session, families will receive tablets with data plans and with the Zoom. They will receive a welcome pack that includes baby gifts that are used to support each session. Dyads in the EHS-CTB digital only group will receive EHS early education, as well as EHS home visitation, and will have access to the CTB content via the CTB App, but will receive no CTB sessions. Content includes videos of baby Elmo and his father and suggested activities.
Who Masked: Outcomes Assessor
Masking Description: Families will be randomly assigned to the treatment or control condition upon enrollment in the study. Because it is an intervention, administered by facilitators, the facilitators and parents will be aware of the treatment families status. The investigators will know which families are receiving the treatment or not because they will need to manage the progress of the intervention and the progress of data collection. Those blind to treatment status will be the data collectors, who will administer all parent surveys and objective measures, including the videotaped parent-child interactions. The coders of the videotaped parent-child interactions will also be blind to treatment status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EHS-CTB Hybrid (Experimental): Dyads in the EHS-CTB hybrid condition will receive 6 individual sessions of CTB conducted by trained facilitators. The first session would be at the center, the 2nd through 5th would be remote, and 6th would be at the EHS center as a group session with other families. Sessions will occur approximately one to two weeks apart, allowing for program completion within 10 weeks. During the first in-person session, families will receive tablets with data plans and with the Zoom. They will receive a welcome pack that includes baby gifts that are used to support each session.
  Interventions: Behavioral: Connect to Baby
- EHS-CTB Digital Only (No Intervention): Dyads in the EHS-CTB digital only group will receive EHS early education, as well as EHS home visitation, and will have access to the CTB content via text messages, but will receive no CTB sessions. Digital content includes videos of Baby Elmo and his father and suggested activities.

INTERVENTIONS:
Behavioral: Connect to Baby — To engage both fathers and mothers, CTB recruits parents at the time of birth, capitalizing on the "magic moment" of delivery, and uses father-inclusive digital media content to engage men. A key innovation lies in the introduction and rehearsal of four interaction skills -- Noticing, Following, Talking, and Encouraging (NiFTE, pronounced "Nifty") -- to foster serve-and-return interactions with infants as well as supportive, cooperative coparenting interactions between mothers and fathers. To maximize program uptake, CTB is situated within an early education program parents already trust and attend. Additionally, the study will test hybrid program delivery with both in-person and remote sessions using video-enabled tablets to reduce scheduling and logistical barriers and thereby enhance retention.
  Arms: EHS-CTB Hybrid

SUMMARY:
The proposed project is a randomized control trial to assess a novel 6-session parenting and coparenting intervention for low-income parents of infants. Connect to Baby (CTB) will be implemented within one of the largest federally-funded early care and education programs, Early Head Start (EHS), in Washington, DC. To engage both fathers and mothers, CTB recruits parents at the time of birth, capitalizing on the "magic moment" of delivery, and uses father-inclusive digital media content to engage men. A key innovation lies in the introduction and rehearsal of four interaction skills -- Noticing, Following, Talking, and Encouraging (NiFTE, pronounced "Nifty") -- to foster serve-and-return interactions with infants as well as supportive, cooperative coparenting interactions between mothers and fathers. To maximize program uptake, CTB is situated within an early education program parents already trust and attend. Additionally, the study will test hybrid program delivery with both in-person and remote sessions using video-enabled tablets to reduce scheduling and logistical barriers and thereby enhance retention. The specific aims of the project are to assess efficacy of random assignment to Hybrid delivery of CTB relative to EHS as usual at enhancing parenting and coparenting quality and parent and child wellbeing. If demonstrated to be efficacious, this program will provide Early Head Start (and other family-serving agencies) a brief cost-effective, manualized preventive intervention that could be used alone or in conjunction with other services to improve parent functioning and co-parenting, further engage fathers in programming and caregiving, and, ultimately, enhance child development.

DETAILED DESCRIPTION:
Overview:

The proposed project is a randomized control trial to assess the effectiveness of a novel 6-session parenting and coparenting intervention for low-income parents of infants designed by the program developers of Just Beginning (JB) and Family Foundations (FF). Connect to Baby (CTB) blends and builds upon these two evidence-based programs and will be implemented within one of the largest federally-funded early care and education programs, Early Head Start (EHS), in Washington, DC. CTB's approach recognizes that although many existing interventions aim to increase parenting quality in low-income contexts, the vast majority yield only modest effects that often fade. These mixed findings stem, in part, from three key weaknesses in existing programs: 1) a focus on mothers, rather than mothers and fathers; 2) a focus on the parent-child relationship to the exclusion of the coparenting relationship; 3) low program recruitment and retention rates. The co-PIs have successfully piloted a program that addresses these weaknesses and can be easily incorporated into programs like EHS to enhance their effects on parenting, and child development. Specifically, to engage both fathers and mothers, CTB recruits parents at the time of birth, capitalizing on the "magic moment" of delivery, and uses father-inclusive digital media content to engage men. A key innovation lies in the introduction and rehearsal of four interaction skills -- Noticing, Following, Talking, and Encouraging (NiFTE, pronounced "Nifty") -- to foster serve-and-return interactions with infants as well as supportive, cooperative coparenting interactions between mothers and fathers. To maximize program uptake, CTB is situated within an early education program parents already trust and attend. Additionally, the study will test hybrid program delivery with both in-person and remote sessions using video-enabled tablets to reduce scheduling and logistical barriers and thereby enhance retention. CTB has two key targets of intervention - coparenting communication and parenting quality. By enhancing these targets, CTB aims to improve parent mental health, and child socioemotional and language outcomes. The specific aims of the project are to assess efficacy of random assignment to Hybrid delivery of CTB relative to EHS as usual at enhancing program targets and both parent mental health and infant socioemotional and language outcomes. If demonstrated to be efficacious, this program will provide Early Head Start (and other family-serving agencies) a brief cost-effective, manualized preventive intervention that could be used alone or in conjunction with other services to improve parent functioning and co-parenting, further engage fathers in programming and caregiving, and, ultimately, enhance child development.

Families will be randomly assigned to CTB-EHS Hybrid and EHS-digital only conditions. There will be 100 dyads randomly assigned to each condition. The main objective of the study is to test the feasibility of the CTB-Hybrid intervention for enhancing targets of co-parenting and parenting, and outcomes of parent well-being and child language and socioemotional development. The specific aims are:

Aim 1. To assess the efficacy of CTB-Hybrid at improving program targets. One hundred and fifty families will be recruited and randomized to one of two conditions: 1) EHS-CTB Hybrid or 2) EHS-digital with CTB digital content (content delivered via the customized application). CTB is hypothesized to increase coparenting communication quality and parenting quality relative to EHS digital at 3- and 6-months post-random assignment (RA); comparing results at each time point will distinguish immediate from sustained effects of the program. Analyses will include both intent-to-treat (ITT) and treatment-on-the-treated (TOT) analyses to determine the importance of program dosage for program efficacy.

Aim 2. To assess the efficacy of CTB-Hybrid at enhancing secondary program outcomes. CTB will also be assessed with regard to parent mental health (assessed using parent self-report and a short diagnostic interview at 3- and 6-months post (RA), and child socioemotional and language outcomes at 3- and 6-months post RA (assessed using parent-report and objective ratings). In exploratory analyses, parenting and coparenting quality will be tested as mediators and child sex as moderator of effects on secondary outcomes.

Study Site:

13 EHS centers in the Washington DC region.

Recruitment, Screening, Enrollment and Informed Consent:

Participants will be recruited at the EHS centers. Informed consent will be collected remotely via zoom and using REDCAP. Given our experiences during the COVID pandemic we will also collect pre and post measures remotely via zoom. For assessment, EHS-digital only and CTB-hybrid families will pick up a packet from the EHS center that includes a data enabled tablet with a zoom link and links to REDCAP survey links and surveys completed on the tablet and a standard set of toys for the assessment. The materials will be returned to the center after the assessment is complete. Except for the child language measure, MCDI, all measures will be administered at each of the three assessment time points. Mindful of the potential burden of lengthy assessments for this high-risk population, assessments will be administered via two Zoom calls that can be done via mobile phone or tablet separated by one week if needed or requested. Non-proprietary measures will be entered into REDCAP and administered on a tablet or mobile phone.

Study Procedures and Evaluations:

Overall study duration and duration of participant involvement. The intervention is 10 weeks long. Participants will also be involved in a pre-assessment, a post-assessment (3 months post random assignment) and a follow-up (6 months post random assignment)

Retention of Study Subjects:

The hybrid delivery is linked to a trusted service (EHS) and the hybrid delivery allows for flexibility in scheduling.

Fidelity Monitoring:

Each CTB facilitator will participate in a two-day training to learn to use the manual and understand the program's principles and how to effectively use the technology to deliver the content remotely run by the lead CTB facilitator. Once facilitators complete training, the first six sessions each facilitator delivers will be video-recorded, via zoom, for fidelity review. During implementation, every 10th session will be recorded and reviewed for fidelity. The trainer, an LCSW will provide individual and group feedback on the extent to which the facilitator followed the manual and engaged parents effectively. Feedback will be based on video review and a fidelity coding scheme created for CTB in which facilitators are scored for session component completion, and 7 positive engagement, 7 negative engagement criteria, every 30 seconds. Pilot data showed that reliability on the fidelity scheme was high (kappa > .7) as was session fidelity and facilitator quality, with low levels of negative engagement and high levels of positive engagement. Any facilitator not delivering CTB with fidelity will receive a refresher training. Moreover, a clinical supervisor and trainer will be available via phone.

ELIGIBILITY:
Inclusion Criteria:

* Must be a mother, father (or father figure, including same sex parent and grandparent) of an infant who is 2-24 months.
* Must speak and read English or Spanish with sufficient fluency for completion of consent forms and questionnaires and actively participate in the intervention.

Exclusion Criteria:

• Pre-intervention assessment their score on the Woman Abuse Screening Tool (WAST) Interpersonal Violence (IPV) screener (Brown, Lent, Schmidt, & Sas, 2000) indicates sexual or physical abuse.

Ages: 2 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Parent Acceptance/Warmth during parent-child interactions | At baseline (when families are enrolled in the study)
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Acceptance/Warmth during parent-child interactions | 3 months
  Qualitative rating (0-4 scale) as coded from a 25 minute parent-child interaction
Parent Acceptance/Warmth during parent-child interactions | 6 months
  Positive parenting behaviors as coded from a 25 minute parent-child interaction
Parent Descriptive Language during parent-child interactions | At baselined (when families enroll in the study)
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Descriptive Language during parent-child interactions | 3 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Descriptive Language during parent-child interactions | 6 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Follows child's lead during parent-child interactions | At baseline (when families enroll in the study)
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Follows child's lead during parent-child interactions | 3 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Follows child's lead during parent-child interactions | 6 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Extends Child's Focus during parent-child interactions | At baseline (when families enroll in the study
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Extends Child's Focus during parent-child interactions | 3 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent Extends Child's Focus during parent-child interactions | 6 months
  Qualitative rating (0-4 scale) as coded from a 25 minute parent-child interaction
Parent restricts child during parent-child interactions | At baseline (when families enroll in the study)
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent restricts child during parent-child interactions | 3 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent restricts child during parent-child interactions | 6 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent criticizes child during parent-child interactions | At baseline (when families enroll in the study)
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent criticizes child during parent-child interactions | 3 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Parent criticizes child during parent-child interactions | 6 months
  Qualitative rating (0-4 scale) of as coded from a 25 minute parent-child interaction
Coparenting Quality:mother-father pleasure in coparenting | At baseline (when families enroll in the study)
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality:mother-father pleasure in coparenting | 3 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality:mother-father pleasure in coparenting | 6 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: displeasure in coparenting | At baseline (when families enroll in the study)
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: displeasure in coparenting | 3 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: displeasure in coparenting | 6 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: interactiveness | at baseline (when families enroll in the study)
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: interactiveness | 3 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: interactiveness | 6 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: cooperation | At baseline (when families enroll in the study)
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: cooperation | 3 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: cooperation | 6 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: competition | At baseline (when families enroll in the study)
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: competition | 3 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Quality: competition | 6 months
  Qualitative rating scale (1-5) as coded from a 25 minutes mother-father-child interaction
Coparenting Relationship Scale | At baseline (when families enroll in the study)
  Coparenting relationship scale measuring quality of communication, 14 items, scale 1-6.
Coparenting Relationship Scale | 3 months
  Coparenting relationship scale measuring quality of communication, 14 items, scale 1-6.
Coparenting Relationship Scale | 6 months
  Coparenting relationship scale measuring quality of communication, 14 items, scale 1-6.
Father Engagement Scale | At baseline (when families enroll in the study)
  Father Engagement Scale, measuring fathers' engagement in 11 activities with infants, scale 0 - 4
Father Engagement Scale | 3 months
  Father Engagement Scale, measuring fathers' engagement in 11 activities with infants, scale 0 - 4
Father Engagement Scale | 6 months
  Father Engagement Scale, measuring fathers' engagement in 11 activities with infants, scale 0 - 4

SECONDARY OUTCOMES:
Parent mental health | At baseline (when families enroll in the study)
  Center for Epidemiologic Studies Depression Scale Revised, scale to measure parent depression symptoms (10-items), scale 0 - 3
Parent mental health | 3 months
  Center for Epidemiologic Studies Depression Scale Revised, scale to measure parent depression symptoms (10-items), scale 0 - 3
Parent mental health | 6 months
  Center for Epidemiologic Studies Depression Scale Revised, scale to measure parent depression symptoms (10-items), scale 0 - 3
Parent self efficacy | at baseline (when families enroll in the study)
  Parental Sense of Competence Scale, 17 items, scale 1 - 6
Parent self efficacy | 3 months
  Parental Sense of Competence Scale, 17 items, scale 1 - 6
Parent self efficacy | 6 months
  Parental Sense of Competence Scale, 17 items, scale 1 - 6
Child language development | At baseline (when families enroll in the study)
  Videotaped parent-infant play task coded using the family interactions using the Individual Growth and Development Indicators (IGDI) Early Communication Indicator (ECI), which codes expressive communication for children between 3 and 36 months.
Child language development | 3 months
  Videotaped parent-infant play task coded using the family interactions using the Individual Growth and Development Indicators (IGDI) Early Communication Indicator (ECI), which codes expressive communication for children between 3 and 36 months.
Child language development | 6 months
  Videotaped parent-infant play task coded using the family interactions using the Individual Growth and Development Indicators (IGDI) Early Communication Indicator (ECI), which codes expressive communication for children between 3 and 36 months.
Child socioemotional development | at baseline (when families enroll in the study)
  The Brief Infant Toddler Social Emotional Assessment (BITSEA), which assesses behavior problems and competencies, 42 items, scale 0 - 2
Child socioemotional development | 3 months
  The Brief Infant Toddler Social Emotional Assessment (BITSEA), which assesses behavior problems and competencies, 42 items, scale 0 - 2
Child socioemotional development | 6 months
  The Brief Infant Toddler Social Emotional Assessment (BITSEA), which assesses behavior problems and competencies, 42 items, scale 0 - 2
Parent Generalized Anxiety Scale | At baseline (when families enroll in the study)
  Scale to measure parent anxiety, Generalized Anxiety Scale, 7 items, scale 0 - 3
Parent Generalized Anxiety Scale | 3 months
  Scale to measure parent anxiety, Generalized Anxiety Scale, 7 items, scale 0 - 3
Parent Generalized Anxiety Scale | 6 months
  Scale to measure parent anxiety, Generalized Anxiety Scale, 7 items, scale 0 - 3
Child Language Development | 3 months
  Scale measuring child expressive and receptive language development, MacArthur-Bates Communicative Development Inventories (MCDI) for infants/toddlers, 89-word vocabulary checklist, 0 - 178 (each item has 0 - 2 scale)
Child Language Development | 6 months
  Scale measuring child expressive and receptive language development, MacArthur-Bates Communicative Development Inventories (MCDI) for infants/toddlers, 89-word vocabulary checklist, 0 - 178 (each item has 0 - 2 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ryan, PhD, Principal Investigator — Georgetown University
Locations (1):
- Child Development and Social Policy Lab, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
This application requests support to collect and maintain a database of contact information, pre- and post-random assignment interview and video records for 200 participants and session recordings for 100 participants for supervision and fidelity tracking. Georgetown University Psychology department will serve as the Data Coordinating Center for this project, utilizing the REDCap database system for secure storage and sharing of research data. Video records will be securely stored and shared on Databrary (www.databrary.org), which is a video repository. While video records require explicit permission, deidentified datasets can also be made available in shared volumes on Databrary and on the open science framework https://osf.io/ to increase accessibility to non-clinical researchers.
Supporting Information: Study Protocol
Time Frame: Data will be made available 12 months after the study completion date.
Access Criteria: The deidentified data will be available to any researchers with access to Databrary or OSF.
URL: https://nyu.databrary.org/

REFERENCES:
- [Background] Richeda B, Smith K, Perkins E, et al. Baby Elmo Leads Dads Back to the Nursery: How a Relationship-Based Intervention for Incarcerated Fathers Enhances Father and Child Outcomes. ZERO TO THREE. 2015;35(5):25-35
- [Background] Feinberg ME, Jones DE, Kan ML, Goslin MC. Effects of family foundations on parents and children: 3.5 years after baseline. J Fam Psychol. 2010 Oct;24(5):532-42. doi: 10.1037/a0020837. PMID 20954763
- [Background] Feinberg ME, Jones DE, Hostetler ML, Roettger ME, Paul IM, Ehrenthal DB. Couple-Focused Prevention at the Transition to Parenthood, a Randomized Trial: Effects on Coparenting, Parenting, Family Violence, and Parent and Child Adjustment. Prev Sci. 2016 Aug;17(6):751-64. doi: 10.1007/s11121-016-0674-z. PMID 27334116
- [Background] Barr R, Brito N, Zocca J, Reina S, Rodriguez J, Shauffer C. The Baby Elmo Program: Improving teen father-child interactions within juvenile justice facilities. Children and Youth Services Review. 2011;33(9):1555-1562. doi:10.1016/j.childyouth.2011.03.020
- [Background] Barr R, Morin M, Brito N, Richeda B, Rodriguez J, Shauffer C. Delivering services to incarcerated teen fathers: a pilot intervention to increase the quality of father-infant interactions during visitation. Psychol Serv. 2014 Feb;11(1):10-21. doi: 10.1037/a0034877. Epub 2013 Nov 18. PMID 24246016
- [Background] Feinberg ME, Kan ML. Establishing family foundations: intervention effects on coparenting, parent/infant well-being, and parent-child relations. J Fam Psychol. 2008 Apr;22(2):253-63. doi: 10.1037/0893-3200.22.2.253. PMID 18410212
- [Background] Feinberg ME, Jones DE. Experimental Support for a Family Systems Approach to Child Development: Multiple Mediators of Intervention Effects across the Transition to Parenthood. Couple Family Psychol. 2018 Jun;7(2):63-75. doi: 10.1037/cfp0000100. PMID 30858994

DOCUMENTS (2):
  • Study Protocol (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT06179576/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT06179576/SAP_001.pdf